CLINICAL TRIAL: NCT04960826
Title: dEoxyniValenol as Risk Factor for Inflammatory Bowel Diseases: Human detoxifiCaTion and Impact On intestiNal Microbiota and Homeostasis
Brief Title: Study of an Environmental Risk Factor in Crohn's Disease
Acronym: EVICTION
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_11; 2020-A02380-39 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-07-01; First posted 2021-07-14 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Crohn's disease patients
- Non IBD patients

SUMMARY:
Inflammatory bowel disease (IBD) are lifelong chronic diseases affecting the gastrointestinal tract. The precise etiology and the different actors participating to the pathophysiological process leading to the disease development are still not well understood. A complex interaction between genetics, gut microbiota and environmental factors is thought to trigger the inappropriate mucosal immune response observed in IBD patients. We hypothesize that DON might be an environmental risk factor for IBD.The focus on the human relevance of the gut effects of DON by studying its exposure, metabolism and adverse effects in health and disease focusing on IBD patients

ELIGIBILITY:
Inclusion Criteria:

* Group 1: patients with ileocolic Crohn's disease requiring surgery
* Group 2: Patients requiring ileal and / or colonic surgery for a reason other than Crohn's disease or ulcerative colitis (for example, cancer, polyp or diverticulum).

Exclusion Criteria:

* Vegetarian or vegan patients, celiac disease, gluten sensitivity, eating disorders, people with a particular diet or eating behavior or suffering from obesity or anorexia
* Surgical history: patient having undergone intestinal resection
* Current treatments: patient receiving antibiotic or probiotic treatment within 6 weeks prior to inclusion / patient having taken topical treatment (suppositories or enema of 5ASA or corticosteroids) within 6 weeks prior to inclusion

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Group 1: patients with ileocolic Crohn's disease requiring surgery
  * Group 2: Patients requiring ileal and / or colonic surgery for a reason other than Crohn's disease or ulcerative colitis (for example, cancer, polyp or diverticulum).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Quantification of Deoxynivalenol and its conjugated metabolites by Liquid Chromatography coupled to tandem Mass Spectrometry (LC-MS/MS). | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ZERBIB, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Lille University Hospital, Lille, France